CLINICAL TRIAL: NCT00125554
Title: Double-Blind, Placebo Controlled Trial of Metyrapone as Augmenting Agent in the Treatment of Major Depression
Brief Title: Metyrapone as Additive Treatment in Major Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HH-PSY-ja-007
Record Dates: First submitted 2005-07-29; First posted 2005-08-01 (Estimated); Last update posted 2005-08-12 (Estimated); Status verified 2005-07

CONDITIONS: Major Depressive Disorder
Keywords: Clinical trial; double-blind; randomized placebo-controlled trial; metyrapone; Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Metyrapone

INTERVENTIONS:
Drug: Metyrapone

SUMMARY:
The purpose of this study is to test whether metyrapone is an effective and safe augmenting agent in the treatment of major depression.

DETAILED DESCRIPTION:
The investigators' understanding of the neuroendocrine pathophysiology of depression has made significant progress in recent years, which should help to develop new remedies. Alterations of the hypothalamic-pituitary-adrenocortical (HPA) axis are the most consistent pathological endocrine findings in depression. Hence, attempts have been made to treat depression by directly targeting HPA-axis activity. Currently, three major pathways are investigated:

* Administration of CRH-antagonists;
* Administration of glucocorticoid-receptor-antagonists; and
* Treatment with steroid-synthesis inhibitors like ketoconazole, aminogluthethimide or metyrapone.

The investigators' aim was to conduct the first prospective, randomized, placebo-controlled, double-blind clinical trial of metyrapone as additive treatment in depression. Metyrapone was preferred, since this compound inhibits selectively the 11β-hydroxylase and the 11β-hydroxysteroid dehydrogenase type 1 (11β-HSD-1), thereby exerting direct effects within the central nervous system (CNS). The additive approach was applied because the intended inclusion of severely depressed patients made a pure placebo group ethically challenging. Furthermore, the continuous use of an antidepressant allowed a standardized follow up after the double-blind period.

The hypotheses to be tested were, whether metyrapone exerts potentiating effects during a standard antidepressant therapy and whether an earlier onset-of-action and an improved overall and sustained treatment response can be achieved. Since GR/MR distribution as well as 11β-HSD-1 activities are subject to sexual dimorphism in humans, the sample was prospectively stratified for gender and balanced for treatment with two selected serotonergic antidepressants, allowing further analysis of gender effects and neuroendocrine treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder; single or recurrent according to DSM-IV criteria (296.2 or 296.3)
* A minimum baseline Hamilton score of 18 points on the Hamilton Rating Scale for Depression (HamD; 21-item version)
* Age from 18 to 75 years
* A drug free period of at least 5 days from antidepressants, antipsychotics, mood stabilizers and all other medications except for mild antihypertensive agents
* A negative urinary drug screening diagnosis

Exclusion Criteria:

* A current DSM-IV diagnosis for other axis I psychiatric disorders
* Serious medical conditions, especially those associated with adrenal insufficiency
* Pregnancy, nursing or refusal to use a reliable method of birth control in women.

Participants were randomly assigned to a study group if they met these criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63
Dates: Start 1998-05; Study Completion 2001-07

PRIMARY OUTCOMES:
Two psychometric criteria defined by the number of responders and time to onset-of-action. The number of responders was considered twice after 3 and 5 weeks by defining the treatment response as a 30% and 50% reduction
the course of concentrations of ACTH, cortisol, 11-deoxycortisol and DHEA.

SECONDARY OUTCOMES:
Other psychometric scores, demographic parameters and side effects were considered as secondary variables.

CONTACTS AND LOCATIONS:
Overall Officials: Holger Jahn, MD, Study Director — University Hospital Hamburg-Eppendorf, Germany
Locations (1):
- Dept. of Psychiatry and Psychotherapy, UKE, Hamburg, Hamburg, Germany

REFERENCES:
- [Result] Jahn H, Schick M, Kiefer F, Kellner M, Yassouridis A, Wiedemann K. Metyrapone as additive treatment in major depression: a double-blind and placebo-controlled trial. Arch Gen Psychiatry. 2004 Dec;61(12):1235-44. doi: 10.1001/archpsyc.61.12.1235. PMID 15583115